CLINICAL TRIAL: NCT02209805
Title: Safety and Pharmacokinetics of BIRB 796 BS Tablets Administered Twice Daily Orally (Total Daily Dose 30, 60, and 120 mg) to Healthy Human Subjects for 14 Days. A Double-blind, Placebo-controlled, Parallel Group Study.
Brief Title: Safety and Pharmacokinetics of BIRB 796 BS Tablets Administered to Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.14
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — doramapimod

ARMS (4):
- BIRB 796 BS, low dose (Experimental)
  Interventions: Drug: BIRB 796 BS, low dose
- BIRB 796 BS, high dose (Experimental)
  Interventions: Drug: BIRB 796 BS, high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BIRB 796 BS, medium dose (Experimental)
  Interventions: Drug: BIRB 796 BS, low dose; Drug: BIRB 796 BS, high dose

INTERVENTIONS:
Drug: BIRB 796 BS, low dose
  Arms: BIRB 796 BS, low dose; BIRB 796 BS, medium dose
Drug: BIRB 796 BS, high dose
  Arms: BIRB 796 BS, high dose; BIRB 796 BS, medium dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the safety and pharmacokinetics of BIRB 796 BS tablets administered as multiple daily doses at various dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice and local legislation
* Age >= 18 and <= 45 years
* Broca >= - 20 % and <= + 20%
* Able to communicate well with the investigator and to comply with study requirements
* > 10 elimination half lives present since last use of any investigational drug for that investigational drug
* Laboratory values within a clinically relevant reference range

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, temperature, and EKG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* History of vasculitis (past history of fever, malaise, myalgias, rash, etc.)
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 1 months prior to administration or during trial)
* Smoker
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Use of methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.) < one week prior to administration of study drug
* Blood donation or loss > 400 mL (< 1 month prior to administration or during the trial)
* Excessive physical activities (< 5 days prior to administration or during the trial)
* Following specific laboratory findings: total white blood cell >= 10 x 109/L, C-Reactive Protein >= 4.5 mg/L, gamma-glutamyl-transferase >= 25 U/L, aspartate transaminase >= 16 U/L, alanine transaminase >= 20 U/L any erythrocytes or > 15 mg/dl protein on urine dipstick
* Any EKG value outside of the reference range of clinical relevance including, but not limited to QTcB > 480 ms, PR interval > 240 ms, QRS interval > 110 ms
* History of any familial bleeding disorder
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2001-01; Primary Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant changes in vital signs | up to 21 days
Number of patients with clinically significant changes in laboratory parameters | up to 21 days
Number of patients with abnormal findings in electrocardiogram | up to 21 days
Number of patients with adverse events | up to 24 days

SECONDARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) for several time points | up to 36 hours after dosing
Area under the plasma concentration versus time curve (AUC) for several time points | up to 36 hours after dosing
Time at which maximum plasma concentration occurred over a dosing interval (tmax) | up to 36 hours after dosing
Terminal elimination rate constant (λZ) | up to 36 hours after dosing
Elimination half-life (t1/2) | up to 36 hours after dosing
Mean residence time (MRT) | up to 36 hours after dosing
Apparent oral clearance (CL/F) | up to 36 hours after dosing
Apparent volume of distribution during the terminal elimination phase, divided by F (bioavailability factor) (Vz/F) | up to 36 hours after dosing